CLINICAL TRIAL: NCT00004190
Title: A Phase I(Limited)/Phase II Study of Oxaliplatin (OXAL) and Gemcitabine (GEMZAR) in Patients With Metastatic Pancreatic Carcinoma
Brief Title: Gemcitabine Plus Oxaliplatin in Treating Patients With Refractory Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-984351; CDR0000067431 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-01-21; First posted 2004-05-25 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; duct cell adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + oxaliplatin (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 immediately followed by oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks. Patients achieving stable disease, partial response, or regressive disease continue with therapy. Patients achieving complete response for two consecutive evaluations receive an additional 2 courses of therapy. Phase I (closed as of 7/5/00): Cohorts of 3-6 patients receive escalating doses of gemcitabine and oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Phase II: Patients receive the MTD of gemcitabine and oxaliplatin as in phase I. Patients are followed every 3 months for 1 year, and then every 6 months for 4 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine and oxaliplatin in treating patients who have refractory locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of gemcitabine plus oxaliplatin in patients with refractory metastatic or locally advanced pancreatic cancer (phase I portion of the study closed as of 7/5/00). II. Determine the objective tumor response rate to this combination regimen in this patient population.

OUTLINE: This is a dose escalation and efficacy study. Patients receive gemcitabine IV over 30 minutes on days 1 and 8 immediately followed by oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks. Patients achieving stable disease, partial response, or regressive disease continue with therapy. Patients achieving complete response for two consecutive evaluations receive an additional 2 courses of therapy. Phase I (closed as of 7/5/00): Cohorts of 3-6 patients receive escalating doses of gemcitabine and oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Phase II: Patients receive the MTD of gemcitabine and oxaliplatin as in phase I. Patients are followed every 3 months for 1 year, and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 32-52 patients (12 patients to phase I (phase I closed as of 7/5/00) and 20-40 to phase II) will be accrued for this study within approximately 11-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ductal or undifferentiated primary pancreatic cancer for which no standard curative therapy exists Progressive locally advanced disease after combined chemotherapy and radiotherapy OR Not a candidate for combined therapy OR Metastatic disease No islet cell, acinar cell, or cystadenocarcinomas Measurable or evaluable disease No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than ULN OR Creatinine clearance at least 60 mL/min Cardiovascular: No symptomatic congestive heart failure No unstable angina No cardiac arrhythmia Other: No other uncontrolled illness No active infection No allergy to platinum compounds, gemcitabine, or antiemetics No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix No evidence of neuropathy except preexisting grade I or II Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy or immunotherapy No concurrent immunotherapy Chemotherapy: No prior chemotherapy for metastatic disease At least 6 months since prior adjuvant chemotherapy, including cisplatin or gemcitabine, for radiosensitization in locally advanced disease No prior cisplatin or gemcitabine for locally advanced disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to 25% or more of bone marrow No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1999-10; Primary Completion 2003-04 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
overall response rate | Up to 5 years

SECONDARY OUTCOMES:
objective tumor response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Alberts SR, Townley PM, Goldberg RM, Cha SS, Sargent DJ, Moore DF, Krook JE, Pitot HC, Fitch TR, Wiesenfeld M, Mailliard JA. Gemcitabine and oxaliplatin for metastatic pancreatic adenocarcinoma: a North Central Cancer Treatment Group phase II study. Ann Oncol. 2003 Apr;14(4):580-5. doi: 10.1093/annonc/mdg170. PMID 12649105
- [Result] Alberts SR, Townley P, Cha SS, et al.: Oxaliplatin and gemcitabine for patients with pancreatic adenocarcinoma: a North Central Cancer Treatment Group (NCCTG) phase II study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-501, 2002.